CLINICAL TRIAL: NCT07303608
Title: Empowering Clients, Preventing Dropout and Improving Outcomes Through Routine Outcome Monitoring and Systematic Client Feedback in Social Services
Brief Title: Improving Outcomes in Social Services Through Routine Outcome Monitoring and Systematic Client Feedback
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Magnus Johansson, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-00833-01; 2023-01738 (Other Grant/Funding Number: Swedish research council for health, working life and welfare (FORTE))
Record Dates: First submitted 2025-11-26; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Substance Use Disorders; Criminal Behavior; Domestic Violence; Social Care; Family Communication; Family Conflict; Child Behavior Problem; Housing; Everyday Activities
Keywords: Social services; Feedback informed treatment; Systematic client feedback; Routine outcome management
MeSH Terms: conditions — Substance-Related Disorders; Criminal Behavior | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback-informed treatment (FIT) (Experimental): Feedback-informed treatment (FIT) added to treatment as usual. The social workers will use FIT together with the participant at each visit or unit of service (week) The components of FIT is administrating the Outcome Rating Scale at the beginning of session and Session Rating Scale at the end of the session, calculating and interpreting the values (digitally or manually) as well as discussing the results, trying to create a culture of feedback (actively seek and value honest client input).
  Interventions: Behavioral: Feedback informed treatment (FIT); Behavioral: Treatment as usual (TAU)
- Treatment as usual (TAU) (Active Comparator): Treatment as usual at social services without the use of the components in Feedback informed treatment.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Feedback informed treatment (FIT) — Consists of digital or paper tools that systematically collect feedback from the client and presents this to counselor or therapist. However, FIT is more than a collection of measures: an approach, both on the part of the social worker and on the part of the organization, where feedback from the client is actively sought and welcomed, and support of flexibility that interventions can be changed during the treatment period to prevent a negative outcome.
  Other Names: Partners for Change Outcome System (PCOMS); Outcome Rating Scale (ORS); System Rating Scale (SRS)
  Arms: Feedback-informed treatment (FIT)
Behavioral: Treatment as usual (TAU) — Psychosocial support and treatment interventions to help clients in social services with various problems. This can be in the form of individual counselling, social casework, family and network interventions, and similar. These interventions include a variation of cognitive, behavioral, family therapeutic and psychodynamic therapeutic techniques as well as methods for supporting and caring for the client rather than treating specific conditions. The task of social services in Sweden borders to that of psychiatry, addiction care and the correctional system, which are organized on a regional or national level, as opposed to the municipal grounding of social services. Interventions are carried out in the client's environment, in outpatient care and through residential treatment facilities.
  Other Names: Social services psychosocial support and treatment

SUMMARY:
In this project the investigators want to test whether a new method FIT (Feedback informed treatment) can improve the interventions people receive through social services. The FIT method involves regularly providing information about how the client think things are going and what the client thinks about the help and care they receive.

DETAILED DESCRIPTION:
A randomized controlled trial conducted in social services' outpatient care, addiction care and in residential treatment. In addition to direct effects of using FIT (Feedback informed treatment), cost-effectiveness, instrument psychometrics and predictive value will be examined. The project include outcome measures for quality of life, behavior and symptoms which have been selected in collaboration with representatives of the users (social workers and clients). The project will also examine both clients' and social workers' experiences of giving and receiving feedback using FIT, as well as examine factors that influence implementation within social services.

Social services have an ambition to use evidence based practice, but there is a lack of methods that can help social workers and the social service to systematically follow and adapt the interventions based on the clients' situation, context and preferences. FIT is an internationally proven system for doing this. If findings of the current project are positive, it can be spread within social services through an existing network of practitioners and with existing digital tools.

Participating units with experience and interest in FIT will be recruited in collaboration with the Swedish FIT network and with already engaged municipalities and treatment units. The project will ensure that participating social workers have sufficient skills and that their workplace is ready to work with FIT. Clients who are granted treatment at the unit will be asked if they want to be included in a study where they can give feedback on the interventions they receive and help to follow their progress. After baseline, they will be randomized to treatment as usual or treatment with the addition of FIT. To support implementation, the therapists in the FIT group will be offered regular supervision.

ELIGIBILITY:
Inclusion Criteria:

People who have been granted assistance under the Social Services Act at includes centers.

Exclusion Criteria:

* People who do not have sufficient knowledge of Swedish or have impaired cognitive functions that prevent them from using FIT in Swedish, as they cannot benefit from the intervention that the study intends to evaluate the effects of. This is assessed by the respective social service.
* People who receive support and treatment interventions that are not voluntary, i.e. interventions according to the Act on the Compulsory Care of Young People (LVU) or the Act on the Compulsory Care of Drug Abusers (LVM)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Main problem level | Baseline, three months, six months and one year
  The participant choose their main problem area that is addressed in their contact with social servises (Work, employment, finances; School, studies; Alcohol, drugs or gambling; Mental health; Violent behavior or crime; Violence in close relationships; Housing and/or everyday routines; Relationship problems; Other) and rate the problems they have experienced in this area on a visual analog scale (0-100) where a higher number indicate more severe problems.

SECONDARY OUTCOMES:
Days of problem in main area | Baseline, three months, six months and one year
  The participant rate the number of days the last months 0-30 that they have experienced problems in their main problem area.
Secondary problem level | Baseline, three months, six months and one year
  The participant can choose one or two secondary problem areas that is addressed in their contact with social services and rate the problem (0-100) they have experienced in this area. A higher number indicate more severe problems.
Days of problem in secondary area | Baseline, three months, six months and one year
  The participant rate the number of days in the last month (0-30) that they have experienced problems in their secondary problem area.
Clinical outcomes in routine evaluation outcome measure (CORE-OM-8) | Baseline, three months, six months and one year
  Patient reported outcome measures. An 8-item alternative brief measure of psychological distress, based on the shorter CORE-OM-6D for this population. Each item is scored 0-4 (0-26 in total). A higher score indicate more severe problems.
EuroQol Five Dimensions (EQ-5D) | Baseline, three months, six months and one year
  Health questionnaire measuring quality of life in five areas: Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each area is rated 1-5 to form an index. A higher score indicate more severe problems.

OTHER OUTCOMES:
Outcome rating scale (ORS) | during experimental treatment, up to 55 weeks
  Individual (personal well-being), Close relationships (family and friends), Social (work, school, friends) and General (life in general) which are assessed according to four visual analog scales. The ORS is intended to be used several times during treatment or psychotherapy to provide a measure of psychological well-being and treatment progress. The score is 0-40. A lower score indicate more severe problems.
Session Rating Scale (SRS) | during experimental treatment, up to 55 weeks
  A simple, four-item visual analogue scale designed to assess key dimensions of a good therapeutic relationships. The SRS is administered, scored (0-40) and discussed at the end of each session to get real time alliance feedback. A higher score indicate a better therapeutic relationship.
Satisfaction with contact and therapeutic relationship | three months, six months and one year
  Single visual analog scale rating the contact with social worker (0-100) higher indicate a better therapeutic relationship.
Reason for ending treatment | three months, six months and one year
  Two follow-up question about if and why the contact with social services has ended.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Johansson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Linköpings kommun, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
IPD might not be shared because participants are at risk of being identified. Some of the participating social service units are small and may only recruit a small number of participants that could be identified through a combination of demographic variables.